CLINICAL TRIAL: NCT06028620
Title: Can Psychopathy be Prevented? Clinical, Neuroimaging and Genetic Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Feggy Ostrosky Shejet, Head of Neuropsychology and Psychophisiology Laboratory, Universidad Nacional Autonoma de Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A1-S-13501
Record Dates: First submitted 2023-08-23; First posted 2023-09-08 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Psychopathic Personality Trait
Keywords: children maltreatment; neurodevelopmental psychopathy; post-traumatic stress disorder; neuroimaging; brain reorganization
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maltreated children (Experimental): The Maltreated Children group was assessed before and after a psychological intervention using clinical scales (anxiety, depression, post-traumatic stress disorder and Callous unemotional traits) and an emotion paradigm through functional magnetic resonance imaging (fMRI). The psychological intervention implemented with the maltreated group was the Trauma Focused-Cognitive Behavior Therapy.
  For this study, 12 to 16 sessions of 60-90 min each, were implemented once a week for 4 months. 14 out of 15 maltreated children completed the TF-CBT units and one week after that, they underwent the post-treatment assessment.
  Interventions: Behavioral: Trauma Focused-Cognitive Behavior Therapy
- Healthy Control group (No Intervention): This group did not have any records of maltreatment. They were assessed using clinical scales (anxiety, depression, post-traumatic stress disorder and Callous unemotional traits) and an emotion paradigm through functional magnetic resonance imaging (fMRI). Their scores and brain images were compared with the maltreatment group before this group underwent psychological treatment.

INTERVENTIONS:
Behavioral: Trauma Focused-Cognitive Behavior Therapy — TF-CBT consisted of 8 units in which different issues realted to trauma are reviewed. Units are: psychoeducation and parenting skills, relaxation techniques, affective expression and regulation, cognitive coping and processing, trauma narrative and processing, in vivo exposure, co-joint sessions and enhancing safety and future growth.
  Arms: Maltreated children

SUMMARY:
The goal of this clinical trial was to learn about the effect of maltreatment on psychological and brain characteristics in a group of children. The main question it aims to answer are: which are the clinical characteristics of maltreated children before and after a psychological intervention? what changes in brain emotional processing after a psychological intervention? and what is the effect of serotonin transporter variants after a psychological therapy? Participants were assessed before and after intervention with:

* clinical measures of anxiety, depression post-traumatic stress and callous-unemotional traits
* functional neuroimaging techniques to measure brain activity.
* A sample of buccal epithelial cells to obtain information on serotonin transporter.

Researchers will compare maltreated children with a group on non-maltreated children to see if there are differences on psychological characteristics and on brain activity before treatment.

DETAILED DESCRIPTION:
Participants Twenty-five children who suffered child abuse were initially referred by a non-governmental shelter in Mexico City. Children were removed from their homes and placed at the shelter because one or both parents were undergoing judicial processes for various crimes, including child abuse. None of the children had ever received psychological therapy because the shelter did not have a protocol for psychological intervention. After a thorough search for the most appropriate therapy, the TF-CBT was chosen. The information was shared with the shelter administrative board. Once authorities and health professionals at the shelter were informed about the aim of the study, they agreed about the appropriateness of the intervention. A group of trained psychologists would apply the TF-CBT as part of the research protocol. Only children who met the inclusion criteria would participate. Parents or primary caregivers gave their informed written consent for their children to participate in the study. Ethical approval of the study was granted, and the research was performed in accordance with the Code of Ethics of the World Medical Association Declaration of Helsinki.

The final sample consisted of an experimental group of 14 MC which included 4 boys and 10 girls (mean age = 8.77 years old, S.D.=1.83), who had experienced a positive history of different types of trauma, and a control group of 10 HC from the general population who were developing normally and were age-matched to the MC (4 boys and 6 girls) (mean age = 9.57 years old, S.D. = 1.91). They were recruited through an advertisement placed at the Faculty of Psychology, National Autonomous University of Mexico UNAM or by direct referral from parents of previous participants in other studies. All were residents of Mexico City. The study protocol was conducted with the approval of the UNAM Institutional Review Board.

Clinical scales A comprehensive clinical battery was used to assess all participants through the administration of the following assessment tools: The Child Depression Inventory-CDI Spanish version. The Spence Children's Anxiety Scale-SCAS standardized on a sample of Mexican children, the Child PTSD Symptom Scale-CPSS Spanish version, and the Inventory of Callous Unemotional Traits-ICU Spanish version.

Procedure The MC group was assessed before and after the implementation of Trauma Focused-Cognitive Behavior Therapy TF-CBT using clinical scales and an emotion paradigm through functional magnetic resonance imaging fMRI. The HC group was also assessed and scanned twice.

Of the total sample, 14 MC completed the TF-CBT modules and came in for their post-treatment assessment session. In addition, the 10 HC who, according to their parents, had not completed any type of psychological intervention during those 4 months, and still met the inclusion criteria for the initial control group were selected and returned for their post-evaluation session.

ELIGIBILITY:
Inclusion Criteria:

For maltreated children group (MC)

* Ages between 7 to 12 years old
* History of trauma or abuse
* Symptoms of Post traumatic stress disorder
* Symptoms of anxiety

For healthy control (HC)

* Ages between 7 to 12 years old
* No history of trauma or abuse
* Absence or low symptoms of Post Traumatic Stress Disorder
* Absence or low symptoms of anxiety

Exclusion Criteria:

• Any neurodevelopmental, medical condition or risk factor other than maltreatment.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Correlations between brain regions and clinical traits after psychological treatment | 6 months
  Post treatment scores on callous-unemotional traits (possible scores from 0 - to 43), depression (possible scores from 0 to 274, and PTSD (possible scores from 0 - 17) will be correlated with brain activation changes post treatment in regions of interest. Lower scores in clinical scales after treatment means a lower clinical symptom. Brain regios activations will be obtained with a fmri scan. BOLD response will be measured in each brain region.

SECONDARY OUTCOMES:
Clinical differences at pre treatment between maltreatment group and healthy control | 1 month
  Characteristics of clinical traits before treatment in maltreatment and healthy control group.
Clinical improvement after treatment | 6 months
  A Reliable Change Index >1.96 will be obtained fron callous-unemotional, depression and PTSD scales of each participant. This index indicates a significant clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Feggy Ostrosky, Ph.D., Principal Investigator — Facultad de Psicología UNAM
Locations (1):
- Facultad de Psicología UNAM, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any data.

REFERENCES:
- [Background] Admon R, Milad MR, Hendler T. A causal model of post-traumatic stress disorder: disentangling predisposed from acquired neural abnormalities. Trends Cogn Sci. 2013 Jul;17(7):337-47. doi: 10.1016/j.tics.2013.05.005. Epub 2013 Jun 12. PMID 23768722
- [Result] Akiki TJ, Averill CL, Abdallah CG. A Network-Based Neurobiological Model of PTSD: Evidence From Structural and Functional Neuroimaging Studies. Curr Psychiatry Rep. 2017 Sep 19;19(11):81. doi: 10.1007/s11920-017-0840-4. PMID 28924828
- [Result] Blair RJ, Leibenluft E, Pine DS. Conduct disorder and callous-unemotional traits in youth. N Engl J Med. 2014 Dec 4;371(23):2207-16. doi: 10.1056/NEJMra1315612. PMID 25470696
- [Result] Blair, R. J. R., Mitchell, D. G. V., Peschardt, K. S., Colledge, E., Leonard, R. A., Shine, J. H., Murray, L. K., & Perrett, D. I. (2004). Reduced sensitivity to others' fearful expressions in psychopathic individuals. Personality and Individual Differences, 37, 1111-1122. https://doi.org/10.1016/j.paid.2003.10.008
- [Result] Bustos, P., Rincón, P., & Aedo, J. (2009). Validación Preliminar de la Escala Infantil de Síntomas del Trastorno de Estrés Postraumático (Child PTSD Symptom Scale, CPSS) en Niños/as y Adolescentes Víctimas de Violencia Sexual. Psykhe (Santiago), 18(2). https://doi.org/10.4067/S0718-22282009000200008
- [Result] Deblinger E, Mannarino AP, Cohen JA, Runyon MK, Steer RA. Trauma-focused cognitive behavioral therapy for children: impact of the trauma narrative and treatment length. Depress Anxiety. 2011 Jan;28(1):67-75. doi: 10.1002/da.20744. Epub 2010 Sep 9. PMID 20830695
- [Result] Decety, J. (2015). The neural pathways, development and functions of empathy. Current Opinion in Behavioral Sciences, 3, 1-6. https://doi.org/10.1016/j.cobeha.2014.12.001
- [Result] Kimonis ER, Goulter N, Hawes DJ, Wilbur RR, Groer MW. Neuroendocrine factors distinguish juvenile psychopathy variants. Dev Psychobiol. 2017 Mar;59(2):161-173. doi: 10.1002/dev.21473. Epub 2016 Sep 12. PMID 27616728
- [Result] Patriat R, Birn RM, Keding TJ, Herringa RJ. Default-Mode Network Abnormalities in Pediatric Posttraumatic Stress Disorder. J Am Acad Child Adolesc Psychiatry. 2016 Apr;55(4):319-27. doi: 10.1016/j.jaac.2016.01.010. Epub 2016 Feb 4. PMID 27015723
- [Result] Viding E, Fontaine NM, Oliver BR, Plomin R. Negative parental discipline, conduct problems and callous-unemotional traits: monozygotic twin differences study. Br J Psychiatry. 2009 Nov;195(5):414-9. doi: 10.1192/bjp.bp.108.061192. PMID 19880931
- [Result] Weems CF, Russell JD, Neill EL, McCurdy BH. Annual Research Review: Pediatric posttraumatic stress disorder from a neurodevelopmental network perspective. J Child Psychol Psychiatry. 2019 Apr;60(4):395-408. doi: 10.1111/jcpp.12996. Epub 2018 Oct 25. PMID 30357832